CLINICAL TRIAL: NCT07360379
Title: Comparing N-Acetylcysteine (NAC) Versus Alpha-Lipoic Acid (ALA) as Adjuncts for Postoperative Pain Management After Laparoscopic Appendectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Mohamed El Mokadem, Clinical Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HM000209
Record Dates: First submitted 2025-12-27; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic Appendectomy; Pain Management; Anti Oxidative Stress
Keywords: Postoperative pain; Laparoscopic appendectomy; N- acetyl cysteine; Alpha lipoic acid; pain management
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Acetylcysteine; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- N- acetyl cysteine (Active Comparator): Patients of this group will receive 600 mg oral N-acetylcysteine 1-2 hours preoperatively
  Interventions: Dietary Supplement: N Acetyl Cysteine
- Alpha Lipoic acid (Active Comparator): Patients of this group will receive 600 mg oral Alpha lipoic acid 1-2 hours preoperatively
  Interventions: Dietary Supplement: Alpha-Lipoic Acid (ALA)
- Placebo (Placebo Comparator): Matching placebo capsules given at identical intervals.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: N Acetyl Cysteine — 600 mg oral N-acetylcysteine 1-2 hours preoperatively
  Arms: N- acetyl cysteine
Dietary Supplement: Alpha-Lipoic Acid (ALA) — 600 mg oral alpha-lipoic acid 1-2 hours preoperatively.
  Arms: Alpha Lipoic acid
Other: Placebo — Matching placebo capsules given at identical intervals.
  Arms: Placebo

SUMMARY:
Postoperative pain remains a major concern following laparoscopic appendectomy, despite advances in minimally invasive surgery and multimodal analgesia. Inadequate pain control delays recovery, prolongs hospital stay, and increases opioid consumption with associated adverse effects. Therefore, identifying safe adjunct therapies that enhance analgesia and reduce opioid requirements is an important clinical goal.

Oxidative stress and inflammation play a critical role in the development and maintenance of postoperative pain. Surgical trauma induces the generation of reactive oxygen species, which sensitize peripheral nociceptors and enhance central pain transmission.

Antioxidants capable of modulating oxidative stress and inflammatory pathways may therefore offer analgesic benefits beyond conventional analgesics.

N-Acetylcysteine (NAC), a glutathione precursor, has demonstrated anti-inflammatory and analgesic properties in both experimental and clinical settings. It reduces oxidative stress, improves microcirculation, and modulates nociceptive signaling.

Alpha-Lipoic Acid (ALA) is another potent antioxidant that acts as a cofactor in mitochondrial metabolism and has proven efficacy in neuropathic pain conditions. However, its role in acute postoperative pain has not been fully investigated.

To our knowledge, no clinical trial has directly compared NAC and ALA in the perioperative setting, and their effects following laparoscopic appendectomy remain unstudied. This randomized controlled trial aims to evaluate the efficacy and safety of NAC and ALA as adjuncts to standard analgesia, with the goal of estimating their effect on postoperative opioid consumption and pain intensity. The results will provide preliminary data to guide larger definitive studies.

Aim of the study The aim of this study is to evaluate and compare the efficacy and safety of N-acetylcysteine (NAC) and alpha-lipoic acid (ALA) as adjuncts to standard postoperative analgesia in patients undergoing laparoscopic appendectomy. Specifically, the study seeks to determine their effects on postoperative pain intensity, opioid consumption, and recovery profile in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, either sex

  * ASA physical status I-III
  * Undergoing laparoscopic appendectomy
  * Able to provide informed consent and take oral medications postoperatively

Exclusion Criteria:

* Chronic opioid use or chronic pain disorder
* Pregnancy or lactation
* Hepatic or renal impairment
* Known hypersensitivity to NAC or ALA
* Complicated appendicitis requiring open surgery or ICU admission

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | At 2 hours, 6 hours, 12 hours , 24 hours , and 48 hours post-surgery
  Pain intensity: VAS at 2, 6, 12, 24, and 48 hours post-surgery (0 = no pain, 10 = worst pain)

SECONDARY OUTCOMES:
Incidence of Nausea and vomiting | Assessed at 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours post-surgery
  assessed on a 3-point scale (0 = none, 1 = mild, 2 = severe)
Rescue analgesia | in 24 and 48 hours post surgery
  time to first opioid request will be assessed
Occurrence of Adverse effects | Occurrence of adverse effects will be assessed at baseline of the study and at 24 hours and 48 hours post surgery.
  Occurrence of adverse effects like dizziness, headache, rash, or gastrointestinal discomfort will be recorded and graded for severity.
Total opioid use | at baseline of the study and at 24 hours and 48 hours post surgery
  Total opioid use will be assessed throughout the study period

IPD SHARING:
Plan to Share IPD: Undecided